CLINICAL TRIAL: NCT06538051
Title: The Effect of Lying Positions on Hemodynamic Parameters in Intensive Care Patients
Brief Title: The Effect of Lying Position on Hemodynamic Parameters in Patients With Mechanical Ventilated and Spontaneously Breathing.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Sevil Olğun, Adnan Menderes University, Aydin Adnan Menderes University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: position
Record Dates: First submitted 2024-07-01; First posted 2024-08-05 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-06

CONDITIONS: Position Sense Disorders; Hemodynamic Instability
Keywords: Patient position; nurse; Hemodynamic parameter; Intensive care unit
MeSH Terms: conditions — Somatosensory Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- lying positions (Other)
  Interventions: Other: lying positions

INTERVENTIONS:
Other: lying positions — All patients were placed in supine, semi-fowler's and lateral positions, respectively. The effects of positions on hemodynamic parameters were examined.

SUMMARY:
Aim: The study was carried out to examine the effect of lying positions on hemodynamic parameters in patients with mechanical ventilation (MV) and spontaneous breathing.

Material and Methods: The research was carried out semi-experimentally with a single-group posttest design, between November 2021 and May 2022 in the Internal Medicine Intensive Care (ICU) Unit a University Hospital. The study of the sample consisted of 60 patients in the ICU. Data were collected with the patient identification form and the hemodynamic parameters follow-up form. The patients were given different lying positions for 3 days. Hemodynamic parameters were measured and recorded at the 10th minute, 1st hour and 2nd hour after position changes. The measurement results obtained were compared with one-way ANOVA test.

DETAILED DESCRIPTION:
Aim: The study was carried out to examine the effect of lying positions on hemodynamic parameters in patients with mechanical ventilation (MV) and spontaneous breathing.

Material and Methods: The research was carried out semi-experimentally with a single-group posttest design, between the dates of 15.11.2021 and 15.05.2022 in the Internal Medicine Intensive Care (ICU) Unit a University Hospital. Since repeated measurements were planned in the study when determining the sample, A-priori power analysis was performed based on ANOVA repeated measures analysis and the effect size was calculated according to the etasquared value (Abd El-Aziz et al., 2021). Accordingly, the sample of the study was calculated as 34 patients to reach at least 80% power within a 95% confidence interval. The research was completed with a total of 60 patients who were spontaneously breathing (n=30) and mechanically ventilated (n=30). Data were collected with the patient identification form and the hemodynamic parameters follow-up form. Right lateral, semi Fowler's, left lateral and supine positions were applied to the patients every 2 hours between 9 am 5 pm for 3 days and then pulse rate, respiratory rate, systolic blood pressure (SBP), diastolic blood pressure (DBP) and oxygen saturation (SpO₂) were measured at 10th minute, 1st hour and 2nd hour. In data analysis, number, arithmetic mean, standard deviation, chi-square, independent groups t test and one-way ANOVA test were used.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized in intensive care for at least 3 days
* over 18 years of age
* monitored
* spontaneously breathing or connected to a mechanical ventilator,
* conscious or unconscious,
* receiving or not receiving oxygen support,
* with or without a tracheostomy,
* hemoglobin level of 8g/dl.

Exclusion Criteria:

* Patients with movement restrictions
* inotropic/vasopressor and sedative group medications
* body temperature of 38˚C and above
* patients receiving CPAP (Continuous Positive Airway Pressure) treatment

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2022-05-15 (Actual)

PRIMARY OUTCOMES:
Respiratory rate | Measurements were made 3 times a day (10th minute, 1st hour and 2nd hour) for 3 days.
  The patients' respiratory rate were measured and compared separately in the supine semi-fowler's and lateral positions.
oxygen saturation | Measurements were made 3 times a day (10th minute, 1st hour and 2nd hour) for 3 days.
  The patients' oxygen saturation were measured and compared separately in the supine semi-fowler's and lateral positions.
Arterial blood pressure | Measurements were made 3 times a day (10th minute, 1st hour and 2nd hour) for 3 days.
  The patients' arterial blood pressure were measured and compared separately in the supine semi-fowler's and lateral positions.
pulse rate | Measurements were made 3 times a day (10th minute, 1st hour and 2nd hour) for 3 days.
  The patients' pulse rate were measured and compared separately in the supine semi-fowler's and lateral positions.

CONTACTS AND LOCATIONS:
Locations (1):
- Sevil Olğun, Aydin, Turkey (Türkiye)